CLINICAL TRIAL: NCT06531265
Title: Cryotechnique as a Diagnostic and Therapeutic Tool of Endobronchial Tumors: A Prospective Study
Brief Title: Cryotechnique as a Diagnostic and Therapeutic Tool of Endobronchial Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Hend Mohammed Abdelraheem Esmaeel, Associate professor, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-24-06--01PD
Record Dates: First submitted 2024-07-19; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Cryotherapy Effect; Bronchial Neoplasms
Keywords: cryobiopsy; cryotherapy; endobronchial tumors
MeSH Terms: conditions — Bronchial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): Endobronchial cryobiopsy and cryotherapy using flexible bronchoscopy
  Interventions: Procedure: Endobronchial cryobiopsy and cryotherapy using flexible bronchoscopy

INTERVENTIONS:
Procedure: Endobronchial cryobiopsy and cryotherapy using flexible bronchoscopy — Bronchoscopic evaluation of endobronchial lesion with biopsy and cryotherapy for recanalisation

SUMMARY:
This study was to assess the diagnostic yield and the safety of bronchoscopic cryotechniques in the management of endobronchial tumors.

DETAILED DESCRIPTION:
Novel flexible cryoprobes were introduced for tissue sampling during bronchoscopy. Employing this approach, the sample is collected when frozen, with the tissue attached to the frozen end of the probe. This approach enables the retrieval of larger tissue samples from endobronchial lesionsEndobronchial cryotherapy is employed to treat individuals with obstructive central bronchial lung cancers. It has been demonstrated to effectively recanalize obstructed respiratory passages, alleviate symptoms, and improve the quality of life for patients in advanced stagesThis study aimed to assess the effectiveness and safety of using bronchoscopic cryotechniques for diagnosing and treating endobronchial malignancies.

ELIGIBILITY:
Inclusion Criteria:

* patients with radiologically suspected endobronchial masses

Exclusion Criteria:

* Patients with contraindications to bronchoscopy.
* uncorrected coagulopathy (if the international normalized ratio (INR) is more than 1.5).
* severe refractory hypoxemia (even after administering the highest possible dose of oxygen, the partial pressure of oxygen ("PaO2") stays below 70 mm Hg.
* hypoventilation with hypercapnia (type 2 respiratory failure).
* severe pulmonary hypertension > 55 mmHg by echocardiography.
* hemodynamic instability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | within 10 days
  The recording of histopathological diagnosis as revealed by cryobiopsy
Recanalization Success | one day following the procedure
  The measurement of degree of airway recanalization through bronchoscopic evaluation

SECONDARY OUTCOMES:
Degree of dyspnea improvement after the procedure | 2 weeks after the procedure
  Measurement of degree of dyspnea before and after the procedure using Modified medical research counsil scale for dyspnea (mMRC scale)

CONTACTS AND LOCATIONS:
Overall Officials: Sabah Ahmed, PHD, Study Director — Cairo University
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No